CLINICAL TRIAL: NCT02109718
Title: A Randomized Controlled Clinical Trial Comparing The Efficacy and Safety of Open Dressing With Petrolatum Jelly vs. Standard Gauze Dressing With Silver Sulfadiazine in the Treatment of Filipino Adults Aged 18-45 Years Old With Superficial Partial Thickness Burns Less Than or Equal to 10% Total Surface Area Who Are Seen at the Philippine General Hospital Burn Outpatient Clinic
Brief Title: A Trial Comparing the Efficacy and Safety of Open Dressing With Petrolatum Jelly vs. Standard Gauze Dressing With Silver Sulfadiazine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of the Philippines (Other)
Collaborators: Committee on Research Implementation and Development (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SUR-2009-06-11-033
Record Dates: First submitted 2014-03-20; First posted 2014-04-10 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Superficial Partial Thickness Burns
Keywords: Burns; Dressings; Outpatient Management; Petrolatum Jelly; Superficial Partial Thickness Burns; Less than or equal to 10% Total Body Surface Area
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open Dressings with Petrolatum Jelly (Experimental): participants randomized to this arm had their wounds dressed with Open Dressing with Petrolatum Jelly
  Interventions: Drug: Open Dressings with Petrolatum Jelly
- Silver Sulfadiazine Gauze Dressing Group (Active Comparator): Participants randomized to this arm had their wounds dressed with Silver Sulfadiazine Gauze Dressing.
  Interventions: Drug: Silver Sulfadiazine Gauze Dressing Group

INTERVENTIONS:
Drug: Open Dressings with Petrolatum Jelly — participants randomized to this arm had their wounds dressed with a thin layer (1mm) of petrolatum gel applied over the burn wound and instructed to reapply the gel as needed in the event of gel coming off.
  Arms: Open Dressings with Petrolatum Jelly
Drug: Silver Sulfadiazine Gauze Dressing Group — Participants randomized to this arm had their wounds dressed using the standard methods at the Burn Center. An initial layer of fine mesh gauze is applied that is laden with a 2mm layer of silver sulfadiazine cream. This is covered with layers of moist gauze and an outer layer of dry gauze, secured by wrapping with rolled gauze. The dressing extends at least 1 inch beyond the wound edge.
  Arms: Silver Sulfadiazine Gauze Dressing Group

SUMMARY:
The Effectiveness of open dressing with petrolatum jelly in minor burns has not been clearly established. This study determined if the use of open dressings with petrolatum jelly as effective as standard gauze dressing with silver sulfadiazine in treating minor burns in terms of time-to-re-epithelialization, incidence of wound infection,incidence of adverse reactions, and patient acceptance.

Non-extensive superficial partial thickness burns constitute a major proportion of burn injuries. Conventional treatment involves regular changing of absorptive dressings including the application of a topical antimicrobial, commonly silver sulfadiazine. A systematic review has found insufficient evidence to support or refute such antimicrobial prophylaxis. Another review compared silver sulfadiazine dressings with other occlusive and non-antimicrobial dressings and found insufficient evidence to guide practice. Other research has suggested that dressings with petrolatum gel are as effective as silver sulfadiazine. This trial sought to compare the effectiveness of conventional silver sulfadiazine dressings with treatment with petrolatum gel alone.

DETAILED DESCRIPTION:
Patients with superficial partial thickness burns less than 10% Total Body Surface Area were recruited. Patients with burns involving the primary areas (face, hand, groin, joints, feet), previous treatment of the burn wound, previous burn injury to the same area, electrical burns, and patients with inhalation injury were excluded Also excluded were patients with diabetes, known sensitivity or allergy to one of the dressings or their constituents and allergy to NSAIDS, those being treated with systemic steroid medication, and patients with AIDS and AIDS related complex. Participants were then randomized to undergo either open dressings with petrolatum jelly or standard gauze dressings with silver sulfadiazine cream. The number of days to complete re-epithelialization was recorded for each patient. The incidence of wound infection and adverse reactions, notably the occurrence of allergic contact dermatitis was also recorded. The study also assessed both dressings in terms of adherence to the wound bed, ease of dressing removal, pain on application and removal of dressings, time required for dressing change and number of dressing changes in between follow-ups..

A total of 50 participants were recruited. Age, sex, race, health condition, location of burn, % Total Body Surface Area area affected, time lag, causative agent, presence of initial cooling maneuver, medical condition, and associated injuries were similar for petrolatum jelly and silver sulfadiazine groups. There was no significant difference with regard to number of days to re-epithelialization. There was also no significant difference between the two treatment groups with regards to pain experienced during application and removal of the dressings, and the number of dressing changes required in between follow-ups. There was, however, a significant difference between open dressings with petrolatum jelly and silver sulfadiazine gauze dressing in terms of adherence to the wound bed, ease of removal of dressings and time required to change dressings. Open dressings with petrolatum jelly were found to be less adherent, easier to remove, and required less time for dressing change.

Single-center, randomized, controlled clinical trial. Consenting adults 18-45 years old with superficial partial thickness burns less than or equal to 10% total body surface area seen within 24 hours of the injury were randomized to daily dressing either with petrolatum gel without top dressings or conventional silver sulfadiazine treatment with gauze dressings. Primary outcomes were blinded assessment of time to complete re-epithelialization, wound infection or allergic contact dermatitis. Secondary outcomes included assessment of ease, time and pain of dressing changes.

50 patients were recruited and follow up data available for 38. Mean time to re-epithelialization was shorter in the treatment group by more than one day within an overall mean healing time of 7.0 days (p = 0.050). No wound infection or dermatitis was observed in either group. Scores for adherence to the wound, ease of dressing removal and time required to change dressings were significantly better in the petrolatum treatment arm (p < 0.01).

Petrolatum gel without top dressings may be at least as effective as silver sulfadiazine gauze dressings with regard to time to re-epithelialization, and incidence of infection and allergic contact dermatitis. Petrolatum gel appears to be an effective, affordable and widely available alternative in the treatment of minor superficial partial thickness burns in adults.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-45 years old
* Superficial partial thickness burns less than or equal to 10% Total Body Surface Area

Exclusion Criteria:

* Patients with burns involving the primary areas (face, hand, groin, joints, feet)
* Previous treatment of the burn wound
* Previous burn injury to the same area, electrical burn, and patients with inhalation injury
* Patients with diabetes, known sensitivity or allergy to one of the dressings or their constituents and allergy to NSAIDS
* Those being treated with systematic steroid medication
* Patients with AIDS and AIDS related complex

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Number of days to complete re-epithelialization | Participants will be followed up until full re-epithelialization of the wound was noted Time to full re-epithelialization was measured in number of days starting from the day of burn injury. An expected average of up to 2 weeks
  Time to full re-epithelialization. Wound assessment was conducted daily by the principal investigator, who was blinded to treatment allocation, after the dressings of the study participant were completely removed, including residual cream or petrolatum gel. Time to full re-epithelialization was measured in number of days starting from the day of burn injury.
Incidence of wound infection | An expected average of up to 2 weeks
  Wounds were inspected for occurrence of clinical signs of infection, including excessive erythema, edema, pain, purulence, and lymphadenitis (tissue biopsies for microbiologic evaluation were planned in the event of clinical signs of infection) until full re-epithelialization.
Incidence of adverse reactions including allergic contact dermatitis (ACD) | An expected average of up to 2 weeks
  Wounds were inspected for occurrence of ACD (defined as extensive pruritus and a positive patch test) until full re-epithelialization.

SECONDARY OUTCOMES:
Dressing adherence (score) | An expected average of up to 2 weeks
  Adherence was scored using the following scale. Adherence of dressing to the wound bed: 1 = "none" (no adherence); 2 = "minimal" (adherence to <25% of wound bed); 3 = "moderate" (adherence to 26-75% of the wound bed; 4 = "firm" (adherence to >75% of wound bed).
Ease of dressing removal (score) | An expected average of up to 2 weeks
  Ease of removal of dressings was scored using the following scale. Ease of removal of dressing: 1 = "easy"; 2 = "moderate"; 3 = "difficult".
Time taken to change dressing (score) | An expected average of up to 2 weeks
  Time taken to change dressing was categorized as: 1 = 1-5 minutes; 2 = 6-10 minutes; 3 = 11-15 minutes; 4 = 16-20 minutes; 5 = 21-25 minutes; 6 = 26-30 minutes.
Number of dressing changes and reapplications during the day (score) | An expected average of up to 2 weeks
  The reported number of dressing changes within the day from last assessment were categorized as: 1 = 0-2 times; 2 = 3-4 times; 3 = > 4 times.
Pain during dressing changes (score) | An expected average of up to 2 weeks
  Participant-reported pain during removal of dressing was evaluated using a visual analogue scale (VAS) of 0-10.
Pain during removal of dressings (score) | An expected average of up to 2 weeks
  Participant-reported pain while dressing the wound was evaluated using a visual analogue scale (VAS) of 0-10.

CONTACTS AND LOCATIONS:
Locations (1):
- Philippine General Hospital - University of the Philippines Manila, Manila, National Capital Region, Philippines

REFERENCES:
- [Derived] Genuino GA, Baluyut-Angeles KV, Espiritu AP, Lapitan MC, Buckley BS. Topical petrolatum gel alone versus topical silver sulfadiazine with standard gauze dressings for the treatment of superficial partial thickness burns in adults: a randomized controlled trial. Burns. 2014 Nov;40(7):1267-73. doi: 10.1016/j.burns.2014.07.024. Epub 2014 Aug 27. PMID 25172229